

## Protocol for non-interventional studies based on existing data:

| Document Number: | c12696196-01 |
|---|---|
| BI Study Number: | 1160.219 |
| BI Investigational Product(s): | PRADAXA (dabigatran) |
| Title: | Validation of predictors for oral anticoagulant medication choice using EMR data |
| | (Phase 3b of the BI/BWH Pradaxa study program) |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | 02 November 2016 |
| PASS: | No |
| EU PAS register number: | Not available yet |
| Active substance: | Dabigatran etexilate |
| Medicinal product: | Pradaxa |
| Product reference: | EU/1/08/442/001-019 |
| Procedure number: | EMEA/H/C/000829 |
| Joint PASS: | Not applicable |
| Research question and objectives: | The research question is whether select patient characteristics that may be incompletely captured by insurance claims data, differ between dabigatran and warfarin initiators. |
| | Objectives: |
| | 1) Descriptive: To identify select clinical covariates from electronic medical records that might be associated with initiation of oral anticoagulant medications (dabigatran or warfarin) in NVAF patients at risk for stroke and are not usually well captured in the associated claims database |
| | 2) Prediction Rule: To assess how well EMR-based clinical characteristics can be captured on the basis of claims data only |
| | Assess Balance: To assess the potential for unmeasured confounding in dabigatran vs warfarin comparative effectiveness and safety studies based on administrative claims |

## **Boehringer Ingelheim**

**** 

## Protocol for non-interventional studies based on existing data:

BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | databases |
|---|---|
| Country(-ies) of study: | US |
| A 41 | |
| Author: | |
| Marketing authorisation holder(s): | Boehringer Ingelheim |
| MAH contact person: | |
| Date: | 02 November 2016 |
| © 2016 Roehringer Ingelheim Ir | Proprietary confidential information |

© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 1. TABLE OF CONTENTS

| TITLE PAGE | 1 |
|-----------------------------------------|----|
| 1. TABLE OF CONTENTS | 3 |
| 2. LIST OF ABBREVIATIONS | 5 |
| 3. RESPONSIBLE PARTIES | 7 |
| 4. ABSTRACT | 8 |
| 5. AMENDMENTS AND UPDATES | 12 |
| 6. MILESTONES | 13 |
| 7. RATIONALE AND BACKGROUND | 14 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 15 |
| 9. RESEARCH METHODS | |
| 9.1 STUDY DESIGN | 16 |
| 9.2 SETTING | 16 |
| 9.3 VARIABLES | 16 |
| 9.3.1 Exposures | 16 |
| 9.3.2 Outcomes | 16 |
| 9.3.2.1 Primary outcomes | 17 |
| 9.3.2.2 Secondary outcomes | 17 |
| 9.3.2.3 Further outcomes | 17 |
| 9.3.3 Covariates | 20 |
| 9.4 DATA SOURCES | 32 |
| 9.5 STUDY SIZE | 33 |
| 9.6 DATA MANAGEMENT | 34 |
| 9.7 DATA ANALYSIS | 34 |
| 9.7.1 Main analysis | 34 |
| 9.7.2 Further analysis | |
| 9.8 QUALITY CONTROL | 38 |
| 9.9 LIMITATIONS OF THE RESEARCH METHODS | 38 |
| 9.10 OTHER ASPECTS | |
| 9.11 SUBJECTS | 39 |
| 9.11.1 Study group | |
| 9.11.2 EMR-linked subset | |
| 9.12 BIAS | |
| 10. PROTECTION OF HUMAN SUBJECTS | 43 |
| 001 MCC 00 124 PD 01 (4 0) | |

# Protocol for non-interventional studies based on existing data: BI Study Number 1160.219

c12696196-01

| 11. | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 44 |
|------|--------------------------------------------------------------|----|
| 12. | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 45 |
| 13. | REFERENCES | 46 |
| 13. | 1 PUBLISHED REFERENCES | 46 |
| 13.2 | 2 UNPUBLISHED REFERENCES | 47 |
| ANN | NEX 1. LIST OF STAND-ALONE DOCUMENTS | 48 |
| ANN | NEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOLS | 49 |
| ΔΝΝ | JEX 3 ADDITIONAL INFORMATION | 55 |

Protocol for non-interventional studies based on existing d

BI Study Number 1160.219 c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

ACCP American College of Chest Physicians ACEI Angiotensin-converting Enzyme Inhibitor

AES Advanced Encryption Standard

AF Atrial Fibrillation

ALT Serum Alanine Aminotransferase ARB Angiotensin Receptor Blocker

ASCVD Atherosclerotic Cardiovascular Disease

BB Beta Blocker

BI Boehringer Ingelheim BMI Body Mass Index

BWH Brigham and Women's Hospital
CABG Coronary Artery Bypass Graft
CAD Coronary Artery Disease
CCB Calcium Channel Blocker

CHA<sub>2</sub>DS<sub>2</sub>-VASc Congestive Heart Failure, Hypertension, Age > 75, Diabetes

Mellitus, Prior Stroke or Transient Ischemic Attack, Vascular

Disease, Age 65-74, Sex Category

CHADS<sub>2</sub> Congestive Heart Failure, Hypertension, Age> 75, Diabetes Mellitus,

Prior Stroke or Transient Ischemic Attack

CHF Congestive Heart Failure
CI Confidence Interval

CONSORT Consolidated Standards for Reporting Trials

CPT Current Procedural Terminology

Cr Creatinine

DM Diabetes Mellitus

DVT Deep Venous Thromboembolism

Dx Diagnosis

EMR Electronic Medical Records
ESC European Society of Cardiology
GFR Glomerular Filtration Rate

GI Gastrointestinal

H2 Receptor Histamine H2 Receptor

HAS-BLED Hypertension, Abnormal Liver/Renal function, Stroke, Bleeding

history or predisposition, Labile INR, Elderly (Age >65), Drugs-

Alcohol usage

HbA1c Hemoglobin A1C

HCPC Healthcare Common Procedure Coding hdPS High-dimensional Propensity Score

HR Hazard Ratio

ICD-9 International Classification of Diseases, Ninth Revision, Clinical

Modification

ICH Intracerebral Hemorrhage
INR International Normalized Ratio

ITT Intent-To-Treat

IRB Institutional Review Board ISF Investigator Site File

## **Boehringer Ingelheim**

## 

#### Protocol for non-interventional studies based on existing data:

## BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

LDL Low Density Lipoprotein

LOS Length of Stay

MDRD Modification of Diet in Renal Disease

MI Myocardial Infarction
NOAC New Oral Anticoagulant

NSAID Non-steroidal Anti-inflammatory Drug

NVAF Non-valvular Atrial Fibrillation PAD Peripheral Artery Disease

PCI Percutaneous Coronary Intervention

PE Pulmonary Embolism

PGP P-glycoprotein

PPI Proton Pump Inhibitor
PPV Positive Predictive Value

PS Propensity Score

PTCA Percutaneous Transluminal Coronary Angioplasty

PVD Peripheral Vascular Disease

PY Person-Year

RE-LY Randomized Evaluation of Long-Term Anticoagulation Therapy

RR Relative Risk

SAH Subarachnoid Hemorrhage SBP Systolic Blood Pressure SCr Serum Creatinine SD Standard deviation

TIA Transient Ischemic Attack t.i.d. ter in die (3 times a day)

US United States

VTE Venous Thromboembolism



BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished med<br>Pradaxa® (Dabigatran<br>warfarin | | | |
| Name of active ingreed Dabigatran etexilate of | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 02 November 2016 | 1160.219 | 1.0 | |
| Title of study: | Association of select EMR-based covariates with oral anticoagulant medication selection Version and date: Version 1.0, 02 November 2016 | | |
| Rationale and background: | A study of safety/effectiveness of dabigatran is being conducted in health insurer claims databases that may incompletely capture select variables representing covariates. This validation study seeks to ascertain a select set of covariates in electronic medical records (EMRs) linked to a subset of patients within the insurance claims data in order to assess the potential for unmeasured confounding in observational studies based on insurance claims databases only. | | |
| Research question and objectives: | The research question is whether select patient characteristics that may be incompletely captured by insurance claims data differ between dabigatran and warfarin initiators. Objectives: | | |
| | <ol> <li>Descriptive: To identify select clinical covariates from electronic medical records that might be associated with initiation of oral anticoagulant medications (dabigatran or warfarin) in patients with NVAF at risk for stroke and are not usually well captured in the associated claims database.</li> <li>Prediction Rule: To quantify the association between EMR-based clinical characteristics and patterns of insurance claims</li> </ol> | | |

# Protocol for non-interventional studies based on existing data: BI Study Number 1160.219

c12696196-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished med<br>Pradaxa® (Dabigatran<br>warfarin | | | |
| Name of active ingree<br>Dabigatran etexilate or | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 02 November 2016 | 1160.219 | 1.0 | |
| Research question and objectives: | confounding in da | ance: To assess the potential for abigatran vs warfarin comparatived on administrative claims datal | e effectiveness and |
| Study design: | A validation study | y | |
| | Patients from an US health insurance database (electronic medical records) with a recorded diagnosis of atrial fibrillation without evidence of valvular etiology and at risk for stroke who initiate dabigatran or warfarin between October 2010 and December 2014 (This date range corresponds to the available matched cohort date range). Inclusion criteria: • A recorded diagnosis of atrial fibrillation. • Initiation of anticoagulant medication (dabigatran or warfarin). • At least 18 years of age on the date of anticoagulant initiation. • CHA₂DS₂-VASc score ≥ 1 • Presence of electronic medical records (for the EMR-based subset) Exclusion criteria: • Patients with missing or ambiguous age or sex information. • Patients with less than 12 months enrolment preceding the date of anticoagulant initiation. • Patients with a dispensing of any oral anticoagulant during the 12 months preceding the date of anticoagulant initiation | | |
| | | with a nursing home stay during bed dabigatran/warfarin initiators | oaseiine |

## Protocol for non-interventional studies based on existing data:

BI Study Number 1160.219

c12696196-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished med<br>Pradaxa® (Dabigatran<br>warfarin | - | | |
| Name of active ingree<br>Dabigatran etexilate or | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 02 November 2016 | 1160.219 | 1.0 | |
| Variables: | Patient characteris covariates) | stics derived from insurance clain | ms (claims-based |
| | medications with reflected different prior to and include | • | some of which might be<br>ectronic medical records<br>characteristics from |
| | Primary Outcomes Obesity Smoking Alcohol consumption Abnormal renal function Bleeding history or predisposition Renal function (estimated GFR) Serum Creatinine Abnormal liver function | | |
| | <ul><li>History of</li><li>History/du</li><li>Uncontroll</li></ul> | f atrial fibrillation<br>adherence<br>ration of hypertension<br>ed Hypertension (for HAS-BLEI<br>ration of CHF | <b>D</b> ) |

BI Study Number 1160.219

c12696196-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished med<br>Pradaxa® (Dabigatran<br>warfarin | | | |
| Name of active ingreed Dabigatran etexilate of | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 02 November 2016 | 1160.219 | 1.0 | |
| Variables: | <ul><li>HAS-BLE</li><li>Use of anti</li></ul> | D Score<br>iplatelets or NSAIDs (needed for | HAS-BLED) |
| Data sources: | This study will be conducted within MarketScan data linked to electronic medical records. | | |
| Study size: | Study cohort: approximately 15,000 dabigatran initiators PS-matched to 15,000 warfarin initiators EMR-linked subset: approx. 5.5% of the study cohort. | | |
| Data analysis: | <ul> <li>Analyses will describe the presence in the claims data of each EMR-based clinical characteristic among initiators of dabigatran and initiators of warfarin.</li> <li>A prediction algorithm to identify in the claims data each of the EMR-based clinical characteristic will be developed. The prediction algorithm will be estimated using a regression model that uses each of the EMR characteristic as the model outcome and all available claims-based covariates as predictors.</li> <li>Strength of association between each EMR-based covariate and medication choice will guide quantitative assessments of potential confounding of the association between anticoagulant and clinical outcomes.</li> </ul> | | |
| Milestones: | Draft Protocol: So<br>Final Protocol: No<br>Draft Report: July<br>Final Report: Sep | ovember 2016<br>y 2017 | |


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. AMENDMENTS AND UPDATES

None.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6. MILESTONES

| Milestone | Planned Date |
|-------------------------------------|------------------|
| Contract | June 2012 |
| Draft protocol | September 2013 |
| Final protocol | November 2016 |
| Start of data collection | 15 November 2016 |
| End of data collection | 15 May 2017 |
| First draft report | July 2017 |
| Registration in the EU PAS register | November 2016 |
| Final report of study results: | September 2017 |

## Protocol for non-interventional studies based on existing data: BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

A number of new oral anticoagulants are being developed and marketed to replace vitamin K antagonists, one of the most important drugs in modern medicine. [P11-11875] Unlike vitamin K antagonists, these new drugs do not require dose titration involving intensive therapeutic monitoring of prothrombin time to achieve target anticoagulation within a narrow therapeutic range. In Phase III studies, these drugs were found to be therapeutically advantageous or non-inferior over warfarin. In the coming years, as many as six new anticoagulants could be on the market and a lack of valid comparative evidence will hinder prescriber and payor decision-making.

Pharmacoepidemiologic studies based on large administrative claims databases are increasingly utilized for that purpose; however, these data are collected for reasons unrelated to research, and as a result, might not contain sufficient information on important confounders, such as body mass index, smoking, family history, or alcohol consumption, leading to residual confounding. Several approaches have been proposed to address the issue of unmeasured confounding, and internal validation studies, based on additional data obtained for a subset of participants in the main study population is one of them. Such studies offer specific advantages since they are more representative of the main study population and allow application of methods that do not require assumptions about the direction of confounding. [R13-2768]

This protocol is for a validation study conducted within a cohort of patients initiating dabigatran or warfarin during October 2010 – December 2014 time period and matched on propensity score (PS). The study will involve targeted data ascertainment from linked patients for enhanced covariate assessment via extraction from electronic medical records using existing electronic data including pre-defined variables, with the goal of describing the presence of covariates not typically present or insufficiently measured in claims data in dabigatran users as compared to users of warfarin and assessing the potential for confounding in the comparative safety research that will be undertaken in other phases of the study program.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. RESEARCH QUESTION AND OBJECTIVES

The objectives of this study are:

- 1) Descriptive: To identify select clinical covariates from electronic medical records that might be associated with initiation of oral anticoagulant medications (dabigatran or warfarin) in patients with NVAF at risk for stroke and are not usually well captured in the associated claims database.
- 2) Prediction Rule: To quantify the association between EMR-based clinical characteristics and patterns of insurance claims
- 3) Assess Balance: To assess the potential for unmeasured confounding in dabigatran vs warfarin comparative effectiveness and safety studies based on administrative claims databases

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This study represents a form of internal validation study that will involve selection of a patient sample, extraction of medical record data, and analyses that will have implications for potential confounding in comparative studies of dabigatran effect.

This study will be conducted within a cohort of NVAF patients at risk for stroke initiating dabigatran or warfarin during October 2010 – December 2014 time period identified in MarketScan research claims database based on Protocol 1160.207 (Sequential Expansion of Comparative Effectiveness of Oral Anticoagulants).

#### 9.2 SETTING



#### 9.3 VARIABLES

#### 9.3.1 Exposures

The primary exposure is new initiation of warfarin or dabigatran. Initiators are defined as no anticoagulation with *any oral anticoagulant* in the 12 months before the index prescription. Comparison between these two groups of initiators will be made with respect to variables obtained from the EMR among patients who have been matched on the propensity score derived from insurance claims data.

#### 9.3.2 Outcomes

EMR-based clinical characteristics that are typically used as covariates will be treated as outcomes in this validation study. Unless otherwise noted, all of these outcomes will have an indicator for being recorded in EMR (Present, Y/N). Index date is the date of dabigatran or

## **Boehringer Ingelheim**

## Protocol for non-interventional studies based on existing data:

BI Study Number 1160.219

c12696196-01


Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

warfarin initiation. All characteristics will be assessed prior and including the medication initiation date (index date). The characteristics presented in <u>Table 1</u> reflect likely availability in the EMR.

### 9.3.2.1 Primary outcomes

- Obesity
- Smoking
- Alcohol consumption
- Abnormal renal function
- Bleeding history or predisposition
- Renal function (estimated GFR)
- Serum Creatinine
- Abnormal liver function

#### 9.3.2.2 Secondary outcomes

- Duration of atrial fibrillation
- History of adherence
- History/duration of hypertension
- Uncontrolled Hypertension (for HAS-BLED)
- History/duration of CHF
- Prior TIA
- Diabetes
- Hyperlipidemia
- HAS-BLED Score
- Use of antiplatelets or NSAIDs (needed for HAS-BLED)

BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Table 1Outcome definitions

| Outcome | Definition | Present | Categories if present |
|---|---|---|---|
| Primary | | | |
| Obesity | Calculated BMI >30 or recorded "obesity" | Y/N | Obese, not-obese based on note of obesity or recorded BMI>30. |
| Smoking | Any note on smoking | Y/N | Current & past combined and nonsmoker & not noted combined. |
| Alcohol consumption | Any note on alcohol use | Y/N | Alcohol use (any);<br>No use |
| Abnormal renal function | Any note of: Dialysis, renal transplant Serum Creatinine >1.3 mg/dL | Y/N | |
| Bleeding history or predisposition | Any note of: Major bleeding requiring hospitalization or blood transfusion or causing a decrease in hemoglobin level of > 2 g/L | Y/N | |
| Renal function | Estimated GFR closest to index dispensing | Y/N | The value |
| Serum Creatinine | Closest to the index date | Y/N | The value |
| Abnormal liver function | Any note of: Liver disease, cirrhosis, Active hepatitis C Active hepatitis B Active hepatitis A AST/ALT >3X upper limit of normal Absence of any note would be considered as absence of the disease | Y/N | |

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Table 1 (cont'd) Outcome definitions

| Outcome | Definition | Present | Categories if present |
|---|---|---|---|
| | Secondary | | |
| Duration of atrial fibrillation | Years/months prior to initiation of dabigatran/warfarin | Y/N | Number of months prior to index date for the earliest note |
| History of adherence | Any note of patient adherence/lack thereof in EMR | Y/N | Non-adherent<br>Adherent |
| History/duration of hypertension | Any note of: Hypertension SBP >120 mmHg Hypertension drugs | Y/N | Number of months prior to index date for the earliest date |
| Uncontrolled<br>Hypertension (for<br>HASBLED) | SBP >160 mmHg using the most recent information prior to index date | Y/N | |
| History/duration of CHF | Any note of:<br>CHF | Y/N | Number of months prior to index date for the earliest note |
| Prior TIA | Any note of TIA | Y/N | Also, number of months prior to index date if noted |
| Diabetes | Any note of: Diabetes Absence of any note of diabetes will be considered as absence of the disease | Y/N | |
| Hyperlipidemia | Any note of;<br>Hyperlipidemia, dyslipidemia,<br>LDL>130 mg/dl | | |
| HAS Bled Score | As recorded (if recorded) or calculated from EMR data. | Recorded/<br>calculated<br>/none | The value |
| Use of antiplatelets or<br>NSAIDs (needed for<br>HASBLED) | Use of aspirin, clopidogrel, prasugrel, ticagrelor or NSADs (within 1 month or on the index date) | Y/N | |
| INR | Closest to the index date | Y/N | The value |

BI Study Number 1160.219

c12696196-01

Table 2 Components of HAS-BLED bleeding risk score\*

| HAS-BLED item | Points |
|--------------------------------------------------|--------|
| Hypertension (uncontrolled) | 1 |
| Abnormal renal and liver function (1 point each) | 1 or 2 |
| Stroke | 1 |
| Bleeding history or predisposition (anemia) | 1 |
| Labile INR | 1 |
| Elderly | 1 |
| Drugs or alcohol (1 point each) | 1 or 2 |

<sup>\*</sup>HAS-BLED score is calculated by adding the specified points for each of the conditions listed. [R10-6394]



| Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|

| _ | Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|

BI Study Number 1160.219 c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| _ | Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|



#### 9.4 DATA SOURCES



## Protocol for non-interventional studies based on existing data: BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.5 STUDY SIZE

This study will identify covariates that represent potential confounding variables among dabigatran and warfarin users within a sampled population. The ability to identify a covariate and the precision for estimating potential confounding from the covariate will depend on the numbers of patients from whom electronic medical record data is extracted, and features of the covariate itself, such as how certain it is to be recorded in the medical record and whether binary (yes/no) or other.

The PS-matched dabigatran and warfarin initiators during Oct 2010– December 2013 period are approximately 20,000 each. Assuming that 5.5% of this study group will be linked to EMR, the EMR-linked subset up to Dec 2013 will consist of approximately 1100 patients in each exposure group.

The precision of estimated prevalence for a covariate obtained from the EMR depends on the prevalence of the covariate, and the sample size. With 10,000 dabigatran initiators, this study will estimate a patient characteristic that has a 10% prevalence with considerable precision (the 95% confidence interval will be 9.4% to 10.6%) (Table 7). A characteristic not captured in claims, but present in the medical record with a prevalence of 10% to 20% is plausibly a confounding variable and so this table enumerates characteristics with these prevalences. The table has not been extended below 10% since such lower prevalence characteristics have progressively less ability to produce meaningful confounding, so that while the study will have less precision to estimate such a characteristic, validation of the presence for such a low prevalence characteristic becomes unnecessary. At the other end of the range presented in the table, a characteristic with a prevalence above 20% will be identified with even greater precision, so that it also does not need to be depicted in the table.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

 Table 7
 Precision of Estimates for Proportion Measures

| Numerator | Denominator | Prevalence | 95% CI | Precision (s.e.) |
|-----------|-------------|------------|--------------|------------------|
| 10 | 100 | 10% | 4.9%-17.6% | 3.0% |
| 100 | 1,000 | 10% | 8.2%-12.0% | 0.9% |
| 1,000 | 10,000 | 10% | 9.4%-10.6% | 0.3% |
| 10,000 | 100,000 | 10% | 9.8%-10.2% | 0.1% |
| 100,000 | 1,000,000 | 10% | 9.9%- 10.1% | 0.003% |
| 20 | 100 | 20% | 12.7%-29.2% | 4.0% |
| 200 | 1,000 | 20% | 17.6%-22.6% | 1.3% |
| 2,000 | 10,000 | 20% | 19.2%-20.8% | 0.4% |
| 20,000 | 100,000 | 20% | 19.8%-20.2% | 0.1% |
| 200,000 | 1,000,000 | 20% | 19.9%- 20.1% | 0.004% |



#### 9.7 DATA ANALYSIS

#### 9.7.1 Main analysis

#### Representativeness of EMR

We will assess whether the subpopulation with linked EMR data is a representative sample of the full MarketScan cohort of oral anticoagulant medication initiators. In the full MarketScan cohort, the proportion of each exposure group with linked EMR data available will be determined. We will evaluate the claims-based covariates in the linked and non-linked subpopulations, separately by exposure group as well as overall, by examining prevalences

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

for categorical covariates and means and standard deviations for continuous covariates. These data will be summarized as in the example <u>Table 8</u> and will allow us to determine if there are any patient characteristics that are over-represented or under-represented in the EMR subpopulation. If EMR linkage is only available for a subset with considerably different characteristics than the full cohort or among a subset where the propensity score balance is not retained, then further remedies might be applied such as stratification or weighting.

Table 8 Association between claims-based covariates and EMR linkage.

| Claims-based covariate | Dabigatran initiators | | Warfarin initiators | |
|---|---|---|---|---|
| | N= | | N= | |
| | Linked | Not linked | Linked | Not linked |
| Proportion (N) | | | | |
| Age | | | | |
| Age category 18-35 | | | | |
| Age category 36-64 | | | | |
| Age category 65-74 | | | | |
| Age category 75+ | | | | |
| Sex | | | | |

### Objective 1: Descriptive

The analyses for this objective will occur within the subpopulation of individuals with linked EMR data and will focus on describing the EMR-based clinical characteristics for the dabigatran and warfarin initiators. This table will provide an evaluation of the association between the EMR clinical characteristics and initiation of dabigatran or warfarin.

The prevalence of each category for categorical characteristics and the mean and standard deviation for continuous characteristics will be calculated (as shown in the example <u>Table 9</u>). This analysis will aid in identifying EMR characteristics that are unbalanced across exposure groups and are therefore potential unmeasured confounders after PS matching.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 9 EMR clinical characteristics in matched dabigatran and warfarin initiators

| EMR clinical characteristic | Dabigatran<br>initiators | Warfarin<br>initiators |
|---|---|---|
| | N= | N= |
| Smoking | | |
| Alcohol consumption | | |
| Obesity | | |

Note: anticoagulant initiation are based on claims data

We will seek to define variables derived from the EMR in a manner that reduces missingness. Accordingly, most variables will be defined as presence or non-presence in the EMR, which we will take as a proxy of being medically-recognized. For example, if smoking is noted in the medical record, it will be recorded as present, if it is not present, it will be assumed that the patient does not smoke. We will also evaluate the patterns of missing data in the EMR clinical characteristics.

#### Objective 2: Prediction Rule


Objective 3: Potential Unmeasured Confounding Assessment





#### 9.7.2 Further analysis

None defined.

### 9.8 QUALITY CONTROL

All aspects of data analysis will be conducted according to standard procedures of the Division of Pharmacoepidemiology. Programming for this project will be conducted by a primary analyst and validated by a separate analyst (validation analyst). For all data processing and analysis steps, the validation analyst will review the program along with input and output data sets, and for select steps of the project will employ double programming techniques to reduce the potential for programming errors.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

This is a validation study and we are not assessing the association between EMR-based patient characteristics and clinical outcomes.

The source claims data include limitations with respect to certainty of the capture of exposure, covariates, and outcomes. As a comprehensive insurance database, essentially all billable medical services will result in claims for reimbursement, so that the certainty of capture is tied to likelihood of a claim being submitted to the insurer.

Although more information on covariates is captured in EMR, some data will be missing in EMR as well. In addition, information is assessed during routine medical care (not in a standardized way) and some variation in assessment persists but cannot be studied within the scope of the study.

As in any EMR source, there could be potentially small number of dabigatran initiators and they might not represent dabigatran initiators in the general population. In addition, the data sources for this study are commercial US data sources (based on employed people and their dependents), so they tend to over-represent working-age people. The data are supplemented with elderly through patients with certain types of Medicare coverage (Medicare Advantage); however, elderly with Medicare Advantage tend to be healthier and more likely to still be employed as compared to elderly with other types of Medicare. These features of data may further limit the generalizability in that the results will be most generalizable to US people who are employed. [P13-03077, P13-03078]

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.10 OTHER ASPECTS

Funding: Boehringer Ingelheim GmbH

#### 9.11 SUBJECTS

### 9.11.1 Study group

The main cohort will consist of patients with NVAF at risk for stroke initiating warfarin and dabigatran, from October 2010 through December 2014.

#### Inclusion criteria:

- Initiation of an oral anticoagulant is defined by a dispensing of an anticoagulant medication (warfarin or dabigatran) in the source data, with no dispensing of any oral anticoagulant in the prior 12 months. The date of that dispensing will be defined as the index date for that initiation.
- At least one ICD-9 diagnosis code of 427.31 (atrial fibrillation) at any time prior to and including the index date
- At least 12 months (365 days) continuous enrollment, defined as ≤32 days enrollment gap using enrollment and disenrollment dates, preceding the index date
- 18 years of age and older at index date
- CHA<sub>2</sub>DS<sub>2</sub>-VASc score  $\geq 1$

#### Exclusion criteria:

- Patients with a nursing home stay during baseline
- Patients with missing or ambiguous age or sex information.
- Patients with a dispensing of any oral anticoagulant during the 12 months preceding and including the index date
- Patients with documented evidence of valvular disease defined as at least 1 inpatient or outpatient ICD-9 Dx code of [R11-4334]

394.x (diseases of mitral valve)

395.x (diseases of aortic valve)

396.x (diseases of mitral and aortic valve)

397.x (diseases of other endocardial structures)

398.9x (other and unspecified rheumatic heart diseases)

V42.2 (heart valve replaced by transplant)

V43.3 (heart valve replaced by a mechanical device/prosthesis)

OR

ICD-9 procedure code 35.1x (open heart valvuloplasty without replacement), 35.2x (replacement of heart valve) [R03-1232]

ÒΡ

one of the following CPT codes:

33660-33665 (atrioventricular valve repair)

33400-33403 (aortic valve valvuloplasty)

33420-33430 (mitral valve repair/valvuloplasty/replacement)

33460 (valvectomy, tricuspid valve, with cardiopulmonary bypass)

33463-33468 (tricuspid valve repair/valvuloplasty/replacement)

33475 (replacement, pulmonary valve)

# **Boehringer Ingelheim**


# Protocol for non-interventional studies based on existing data:

BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

33496 (prosthetic valve dysfunction repair)

0257T (implantation of catheter-delivered prosthetic aortic heart valve; open thoracic approach)

0258T (transthoracic cardiac exposure for catheter-delivered aortic valve replacement; without cardiopulmonary bypass)

0259T (transthoracic cardiac exposure for catheter-delivered aortic valve replacement; with cardiopulmonary bypass)

0262T (implantation of catheter-delivered prosthetic pulmonary valve, endovascular approach)

at any time prior to and including the index date.

#### Cohort formation

Initiators of dabigatran and warfarin will be matched on their PS to initiate the treatment of interest (dabigatran) and the calendar quarter of initiation. PS will be derived from predicted probabilities of treatment initiation with dabigatran as compared to warfarin estimated in a logistic regression model that includes all claims-based covariates identified in this protocol

The PS will be

used to match dabigatran initiators to warfarin initiators on a 1:1 fixed ratio basis using a nearest-neighbor algorithm.

#### 9.11.2 EMR-linked subset

From the PS-matched cohorts we will identify patients who have EMR data available. Most analyses will be performed in this group. We expect that the EMR-linked subset is a random subset so that the covariate balance achieved by propensity score matching in the overall cohorts will be retained in the EMR subsets. However, due to chance, some imbalances in baseline characteristics may occur. We will check the average PS among the linked subset and inspect covariates among them prior to proceeding with the analysis. In the event of imbalances, we will proceed with analyses outlined after stratifying by the propensity score.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Figure 1 Patient Selection Flow Chart



We will provide Truven with linkage IDs and exposure indicators. Within the EMR-linked subset, Truven will evaluate the balance of the EMR clinical characteristics across exposure groups (see <u>section 9.7 Data Analysis</u> for detailed description).

# Protocol for non-interventional studies based on existing data: BI Study Number 1160.219

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.12 **BIAS**

Various design and analysis methods will be implemented to reduce the potential for bias in the study. We will employ new-user cohorts of dabigatran and warfarin in order to address differences that might arise in the comparison of newer and older treatments, such as survivor bias and attrition of susceptibles. The comparator cohort will be formed warfarin initiators with similar clinical profiles to dabigatran initiators to reduce confounding by indication. We will employ propensity score matching of dabigatran and warfarin cohorts in order to improve the balance of the cohorts with respect to numerous variables.

As a validation study, the aim of this study is to assess the magnitude of potential confounding that might be present in the main cohort study as a result of non-claims characteristics that are both associated with choice of anticoagulant and predictive of study outcomes.

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10. PROTECTION OF HUMAN SUBJECTS

This study will be submitted to the Institutional Review Board (IRB) of

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

As an observational study based on existing data all patient data will be de-identified and analyzed in aggregate. Individual patient safety related information will not be captured during this study. Thus, individual safety reporting is not applicable for this study.

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The interim and final reports will consist of a description of the methods, including patient selection and variable definitions along with tabular summaries of cohort characteristics, numbers of patients receiving each anticoagulant and associated follow-up time. Counts of outcomes and corresponding rates and measures of association will be presented. The tabular results will be followed by an interpretive summary along with a discussion of the findings and implications.

Manuscripts describing this work will be submitted for publication in peer-review journals. Findings may also be submitted for presentation at scientific conferences.

# 13. REFERENCES

### 13.1 PUBLISHED REFERENCES

| P11-11875 | Potpara TS, Lip GY. New anticoagulation drugs for atrial fibrillation. Clin Pharmacol Ther 2011;90:502-6. |
|---|---|
| R13-2768 | Sturmer T, Glynn RJ, Rothman KJ, Avorn J, Schneeweiss S. Adjustments for unmeasured confounders in pharmacoepidemiologic database studies using external information. Med Care 2007;45:S158-65. |
| R11-4334 | Birman-Deych E, Waterman AD, Yan Y, Nilasena DS, Radford MJ, Gage BF. Accuracy of ICD-9-CM codes for identifying cardiovascular and stroke risk factors. Med Care 2005;43:480-5. |
| R03-1232 | Go AS, Hylek EM, Borowsky LH, Phillips KA, Selby JV, Singer DE. Warfarin use among ambulatory patients with nonvalvular atrial fibrillation: the anticoagulation and risk factors in atrial fibrillation (ATRIA) study. Ann Intern Med 1999;131:927-34. |
| P06-10925 | Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation. JAMA 2001;285:2864-70. |
| R10-5332 | Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest 2010;137:263-72. |
| R10-6394 | Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest 2010;138:1093-100. |
| P12-01676 | You JJ, Singer DE, Howard PA, et al. Antithrombotic therapy for atrial fibrillation: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest 2012;141:e531S-75S. |
| R11-4190 | Granger CB, Alexander JH, McMurray JJ, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med 2011;365:981-92. |
| P09-11669 | Connolly SJ, Ezekowitz MD, Yusuf S, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med 2009;361:1139-51. |
| R11-4223 | Patel MR, Mahaffey KW, Garg J, et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med 2011;365:883-91. |

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| - | |
|---|---|
| P14-04526 | Camm AJ, Lip GY, De Caterina R, et al. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: An update of the 2010 ESC Guidelines for the management of atrial fibrillation * Developed with the special contribution of the European Heart Rhythm Association. Europace 2012;14:1385-413. |
| R13-4176 | Olesen JB, Lip GY, Hansen PR, et al. Bleeding risk in 'real world' patients with atrial fibrillation: comparison of two established bleeding prediction schemes in a nationwide cohort. J Thromb Haemost 2011;9:1460-7. |
| R13-0521 | Molnar AO, Coca SG, Devereaux PJ, et al. Statin use associates with a lower incidence of acute kidney injury after major elective surgery. J Am Soc Nephrol 2011;22:939-46. |
| R11-4329 | Winkelmayer WC, Schneeweiss S, Mogun H, Patrick AR, Avorn J, Solomon DH. Identification of individuals with CKD from Medicare claims data: a validation study. Am J Kidney Dis 2005;46:225-32. |
| P12-05791 | FDA draft guidance for industry on Drug Interaction Studies - Study Design, Data Analysis, and Implications for Dosing and Labelling. Feb 2012. |
| R12-0541 | Friberg L, Rosenqvist M, Lip GY. Evaluation of risk stratification schemes for ischaemic stroke and bleeding in 182 678 patients with atrial fibrillation: the Swedish Atrial Fibrillation cohort study. Eur Heart J 2012;33:1500-10. |
| P13-03077 | West SL, Strom BL, Freundlich B, Normand E, Koch G, Savitz DA. Completeness of prescription recording in outpatient medical records from a health maintenance organization. J Clin Epidemiol 1994;47:165-71. |
| P13-03078 | West SL, Savitz DA, Koch G, Strom BL, Guess HA, Hartzema A. Recall accuracy for prescription medications: self-report compared with database information. Am J Epidemiol 1995;142:1103-12. |

# 13.2 UNPUBLISHED REFERENCES

None

c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

None

Protocol for non-interventional studies based on existing data:

BI Study Number 1160.219

c12696196-01









c12696196-01





c12696196-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **ANNEX 3. ADDITIONAL INFORMATION**

None